CLINICAL TRIAL: NCT04809792
Title: Magnetic Resonance Imaging-Guided Radiotherapy for Head & Neck SBRT on the 1.5T MR-Linac
Brief Title: MR-Linac for Head and Neck SBRT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Irene Karam, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1509
Record Dates: First submitted 2021-03-15; First posted 2021-03-22 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer
Keywords: Adaptive radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Head and neck cancer (Experimental): In this arm patients with head and neck cancers treated with SBRT are recruited.
  Interventions: Radiation: SBRT on the MR-Linac

INTERVENTIONS:
Radiation: SBRT on the MR-Linac — Radiotherapy is performed on the 1.5 T MR Linac

SUMMARY:
This study will evaluate the feasibility and safety of using MR-guided adaptive Head and Neck stereotactic radiotherapy (SBRT) at each fraction on the 1.5T MR-Linac.

DETAILED DESCRIPTION:
At the Sunnybrook Odette Cancer Centre (OCC), stereotactic body radiation therapy (SBRT) (35- 50 Gy in 5 fractions delivered 2x/week) has been employed in a subgroup of palliative Head and Neck cancer (HNC) patients, as part of an institutional protocol, when greater tumor response is desirable when compared to more palliative regimens.

The MR-Linac has been approved by Health Canada for radiation treatment. With superior soft tissue contrast and the possibility for daily plan adaptation, it allows for higher treatment precision delivery, improved target coverage and greater normal tissue sparing.

As a first step, this study will evaluate the feasibility and safety of using the 1.5T MR-Linac on patients with HNC who are treated with SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Karnofsky performance status score of ≥70
* Biopsy-proven oligometastatic cancer to the HN
* Biopsy-proven primary HN cancer (either mucosal, nodal, skin)
* Patients deemed unsuitable by the treating radiation oncologist for radiation treatment with curative intent owing to advanced age, significant comorbidities, poor performance status, distant metastatic disease.
* ≥ 1 site amenable to HN SBRT
* Capable of providing informed consent
* Required to complete any systemic therapy ≥ 10 days prior to planned start of HN SBRT, with no plans to initiate systemic therapy ≥10 days following completion of HN SBRT.

Exclusion Criteria:

* History of radiation within the projected treatment field
* Contraindications to MR imaging per institutional policy
* Patients with connective tissue disorders
* History of severe claustrophobia
* Pregnant and or breastfeeding females
* Having an estimated glomerular filtration rate (GFR) <40 ml/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who complete ≥80% of treatment fractions in ≤60 minutes. | 2 years
  Clinical feasibility of delivering radiotherapy treatment on the MR Linac within 60 minutes and the need for patients to transfer to a CT-based linear accelerator will be monitored. The radiotherapy timing sheet will be used to record the length of time for patients to have their MR guided adaptive radiotherapy for each fraction.

SECONDARY OUTCOMES:
Dosimetric outcomes in HN SBRT patients treated with MR-guided adaptation as compared to non-adaptive HN SBRT. | 2 years
  Prospectively recorded OAR dose, cumulative GTV/PTV dose, and projected dose that would have been delivered by non-adaptive plans.
Number of participants with Acute and Late Toxicity | 2 years
  Acute toxicity (during and up to 3 months from the end of treatment) and late toxicity (after 3 months) secondary to SBRT will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0) scale.
Quality of Life as measured by the MD Anderson Symptom Inventory - Head and Neck (MDASI-HN) | 2 years
  Patient Reported Outcome (PRO) measure of symptoms
Quality of Life as measured by the MD Anderson Dysphagia Inventory (MDADI) | 2 years
  Patient Reported Outcome (PRO) measure of symptoms
Quality of Life as measured by the Xerostomia Questionnaire (XQ) | 2 years
  Patient Reported Outcome (PRO) measure of symptoms
Quality of Life as measured by the Patient experience Questionnaire for MR-Linac | 2 years
  Patient Reported Outcome (PRO) measure of symptoms
Locoregional control 6 months based on RECIST criteria 1.1 and assessed on MRI or CT scan imaging | 6 months
  Calculated from time of treatment completion to disease progression at primary site or regional lymph nodes
Progression-free survival | 2 years
  Calculated as time from diagnosis to either death or detection of recurrent disease
Overall survival | 2 years
  Calculated as time from diagnosis to either death or last follow-up
Changes in tumor apparent diffusion coefficient (ADC) maps from diffusion weighted (DWI) MRI scan at baseline and at each fraction | 2 years
  Functional imaging kinetics as a correlate of treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Irene Karam, Principal Investigator — Sunnybrook Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No